CLINICAL TRIAL: NCT04383210
Title: CRESTONE: A Phase 2 Study of Seribantumab in Adult Patients With Neuregulin-1 (NRG1) Fusion Positive Locally Advanced or Metastatic Solid Tumors
Brief Title: Study of Seribantumab in Adult Patients With NRG1 Gene Fusion Positive Advanced Solid Tumors
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Business decision
Sponsor: Elevation Oncology (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ELVCAP-001-01
Record Dates: First submitted 2020-05-07; First posted 2020-05-12 (Actual); Results first posted 2025-04-03 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Locally Advanced Solid Tumor; Metastatic Solid Tumor; Pancreatic Cancer; Lung Cancer; Head and Neck Cancer; Breast Cancer; Kidney Cancer; Colorectal Cancer; Bladder Cancer; Ovarian Cancer; Sarcoma; Gallbladder Cancer; Bile Duct Cancer; Esophageal Cancer; Uterine Cancer; Cholangiocarcinoma; Prostate Cancer
Keywords: NRG1; Neuregulin 1; Gene fusion
MeSH Terms: conditions — Neoplasm Metastasis; Pancreatic Neoplasms; Lung Neoplasms; Head and Neck Neoplasms; Breast Neoplasms; Kidney Neoplasms; Colorectal Neoplasms; Urinary Bladder Neoplasms; Ovarian Neoplasms; Sarcoma; Gallbladder Neoplasms; Bile Duct Neoplasms; Esophageal Neoplasms; Uterine Neoplasms; Cholangiocarcinoma; Prostatic Neoplasms; Fibromatosis, Gingival, 2 | interventions — seribantumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cohort 1 (Experimental): A minimum of 55 adult advanced solid tumor patients harboring NRG1 gene fusions, who have received prior standard treatment, excluding prior ERBB-directed therapy.
  Seribantumab 1-h IV infusion at various doses once weekly, every 2 weeks and every 3 weeks, during the induction, consolidation and maintenance dosing phases, respectively.
  Interventions: Drug: Seribantumab
- Cohort 2 (Experimental): Up to 10 adult advanced solid tumor patients harboring NRG1 gene fusions, who have received prior standard treatment, including prior ERBB-directed therapy.
  Seribantumab 1-h IV infusion at various doses once weekly, every 2 weeks and every 3 weeks, during the induction, consolidation and maintenance dosing phases, respectively.
  Interventions: Drug: Seribantumab
- Cohort 3 (Experimental): Up to 10 adult advanced solid tumor patients harboring NRG1 gene fusions lacking an EGF-like domain, who have received prior standard treatment, which may have included prior ERBB-directed therapy.
  Seribantumab 1-h IV infusion at various doses once weekly, every 2 weeks and every 3 weeks, during the induction, consolidation and maintenance dosing phases, respectively.
  Interventions: Drug: Seribantumab

INTERVENTIONS:
Drug: Seribantumab — Anti-HER3 monoclonal antibody

SUMMARY:
This study is an open-label, international, multi-center, Phase 2 study in adult patients with recurrent, locally-advanced or metastatic solid tumors, which harbor the NRG1 gene fusion.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for participation in the study, patients must meet the following inclusion criteria:

* Locally-advanced or metastatic solid tumor with an NRG1 gene fusion identified through molecular assays, such as PCR, NGS (RNA or DNA) or FISH, by a CLIA-certified or similarly accredited laboratory
* Availability of fresh or archived FFPE tumor sample to be submitted to a central laboratory for confirmation of NRG1 gene fusion status
* Patients should have received a minimum of one prior standard therapy appropriate for their tumor type and stage of disease, progressed or been nonresponsive to these available therapies, with no further available curative therapy options
* ≥ 18 years of age
* ECOG performance status (PS) 0, 1 or 2
* Patients must have at least one measurable extra-cranial lesion as defined by RECIST v1.1
* Adequate hepatic function defined as:
* Serum AST and serum ALT < 2.5 × upper limit of normal (ULN), or AST and ALT < 5 × ULN if liver function abnormalities due to underlying malignancy
* Total bilirubin < 2.0 ULN. Subjects with a known history of Gilberts Disease and an isolated elevation of indirect bilirubin are eligible
* Adequate hematologic status, defined as:
* Absolute neutrophil count (ANC) ≥1.5 × 109/L not requiring growth factor support for at least 7 days prior to Screening, and
* Platelet count ≥100.0×109/L not requiring transfusion support for at least 7 days prior to Screening
* Able to provide informed consent or have a legal representative able and willing to do so
* Ability to comply with outpatient treatment, laboratory monitoring, and required clinic visits for the duration of study participation
* Willingness of men and women of reproductive potential to observe conventional and effective birth control for the duration of treatment and for 3 months following study completion; this may include barrier methods such as condom or diaphragm with spermicidal gel.

Exclusion Criteria:

* Known, actionable oncogenic driver mutation other than NRG1 fusion where available standard therapy is indicated
* Life expectancy < 3 months
* Pregnant or lactating
* Prior treatment with ERBB3/HER3 directed therapy (Cohort 1 only)
* Prior treatment with pan-ERBB or any ERBB/HER2/HER3 directed therapy (Cohort 1 only)
* Symptomatic or untreated brain metastases (Note: Patients with asymptomatic brain metastases treated with radiation or surgery and without evidence of progression by imaging at screening are eligible to participate in the study. Patients requiring ongoing corticosteroids to treat brain metastases will not be eligible).
* Received other investigational agent or anticancer therapy within 28 days prior to planned start of seribantumab or 5 half-lives, whichever is shorter
* Prior to initiation of seribantumab treatment, patients must have recovered from clinically significant toxicities from prior anticancer or investigational therapy
* Any other active malignancy requiring systemic therapy
* Known hypersensitivity to any of the components of seribantumab or previous CTCAE grade 3 or higher hypersensitivity reactions to fully human monoclonal antibodies
* Clinically significant cardiac disease, including symptomatic congestive heart failure, unstable angina, acute myocardial infarction within 12 months of planned first dose, or unstable cardiac arrhythmia requiring therapy (including torsades de pointes)
* Active uncontrolled systemic bacterial, viral, or fungal infection
* Patients who are not appropriate candidates for participation in this clinical study for any other reason as deemed by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2020-09-29 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-02-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (42):
- United States (35):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - HonorHealth, Scottsdale, Arizona
  - Compassionate Care Research Group Inc., Fountain Valley, California
  - Pacific Shores Medical Group, Huntington Beach, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of California - Irvine Medical Center, Orange, California
  - University of Colorado Denver, Denver, Colorado
  - Medical Oncology Hematology Consultants, Newark, Delaware
  - Georgetown University, Washington D.C., District of Columbia
  - Moffitt Cancer Center, Tampa, Florida
  - University Cancer And Blood Center, Athens, Georgia
  - Hawaii Cancer Care, Honolulu, Hawaii
  - Northwestern University, Chicago, Illinois
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Henry Ford, Detroit, Michigan
  - Metro Minnesota CCOP, Saint Louis Park, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - The Ohio State University, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Penn State Health Hershey Medical Center Cancer Institute, Hershey, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Sanford Oncology Clinic, Sioux Falls, South Dakota
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Texas Oncology-Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - The University of Texas M.D. Anderson Cancer Center, Houston, Texas
  - Utah Cancer Specialists, Salt Lake City, Utah
  - Oncology & Hematology Associates of Southwest Virginia Inc., DBA Blue Ridge Cancer Care, Blacksburg, Virginia
  - Virginia Cancer Specialists, Fairfax, Virginia
  - Northwest Medical Specialties, PLLC, Tacoma, Washington
  - ThedaCare Regional Cancer Center, Appleton, Wisconsin
  - University of Wisconsin, Madison, Wisconsin
- Australia (4):
  - St. Vincent's Hospital, Sydney, New South Wales
  - Royal Hobart Hospital, Hobart, Tasmania
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Linear Clinical Research Ltd., Nedlands, Western Australia
- Canada (2):
  - BC Cancer, Vancouver, British Columbia
  - William Osler Health System, Brampton, Ontario
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Patil T, Lin JJ, Cheema PK, Carrizosa DR, Burkard ME, Elamin YY, Desai J, Patel JD, Nagasaka M, Reckamp KL, Waqar SN, Bauman JR, Schram AM, Gadgeel SM, Ma PC, Konduri K, Nguyen D, Misleh J, Bleeker J, Weiss M, Thavaneswaran S, Haura EB, Deegan M, Kaufman J, Srivastava J, Jansen VM, Liu SV. CRESTONE: A Phase II Study of the Efficacy and Safety of the HER3 Monoclonal Antibody, Seribantumab, in Solid Tumors With Neuregulin-1 (NRG1) Fusions. JCO Precis Oncol. 2025 Aug;9:e2500221. doi: 10.1200/PO-25-00221. Epub 2025 Dec 22. PMID 41428976

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: Enrolled 36 adult advanced solid tumor patients harboring NRG1 gene fusions, who have received prior standard treatment, excluding prior ERBB-directed therapy.
  Seribantumab 1-h IV infusion at various doses once weekly, every 2 weeks and every 3 weeks, during the induction, consolidation and maintenance dosing phases, respectively.
  Seribantumab: Anti-HER3 monoclonal antibody
- Cohort 2: Enrolled 11 adult advanced solid tumor patients harboring NRG1 gene fusions, who have received prior standard treatment, including prior ERBB-directed therapy.
  Seribantumab 1-h IV infusion at various doses once weekly, every 2 weeks and every 3 weeks, during the induction, consolidation and maintenance dosing phases, respectively.
  Seribantumab: Anti-HER3 monoclonal antibody
- Cohort 3: Enrolled 7 adult advanced solid tumor patients harboring NRG1 gene fusions lacking an EGF-like domain, who have received prior standard treatment, which may have included prior ERBB-directed therapy.
  Seribantumab 1-h IV infusion at various doses once weekly, every 2 weeks and every 3 weeks, during the induction, consolidation and maintenance dosing phases, respectively.
  Seribantumab: Anti-HER3 monoclonal antibody
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Started | 36 | 11 | 7
Completed | 36 | 11 | 7
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Total
Number analyzed (Participants) | 36 | 11 | 7 | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 21 | 6 | 3 | 30
  >=65 years | 15 | 5 | 4 | 24
Age, Continuous [Median (Full Range); unit: years] | 61 [38 to 80] | 59 [19 to 84] | 66 [57 to 72] | 62 [19 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 7 | 5 | 34
  Male | 14 | 4 | 2 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 4 | 4 | 0 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 5 | 0 | 0 | 5
  White | 26 | 6 | 7 | 39
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Canada | 2 | 2 | 0 | 4
  United States | 32 | 9 | 6 | 47
  Australia | 2 | 0 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Description: Tumor assessments were evaluated at baseline by computerized tomography (CT) or magnetic resonance imaging (MRI). The primary objective of this study was to determine the overall objective response rate (ORR) per investigator assessment, defined as confirmed complete response (CR; disappearance of all target lesions) + partial response (PR; at least a 30% decrease in the sum of the longest diameter of target lesions) by RECIST v1.1, for seribantumab monotherapy (3,000 mg QW) in patients with centrally confirmed NRG1 fusion.
Time Frame: Up to 12 months
Population: Among the 36 patients enrolled in Cohort 1, 29 of 36 patients met criteria (criteria includes centrally confirmed NRG1 fusion status and patient received 3,000 mg QW dosing) to be included in the primary efficacy population and were evaluable for investigator assessed response per RECIST v1.1. In Cohorts 2 and 3, one patient in each cohort was not evaluable for investigator assessed response per RECIST v1.1.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 29 | 10 | 6
Participants | 10 | 1 | 0

ADVERSE EVENTS:
Time Frame: 3 years, 4 months
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
All-Cause Mortality (participants affected / at risk) | 21/36 | 8/11 | 7/7
Serious Adverse Events (participants affected / at risk) | 17/36 | 6/11 | 4/7
Other Adverse Events (participants affected / at risk) | 35/36 | 11/11 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=36) | Cohort 2 (N=11) | Cohort 3 (N=7)
Pneumonia (Infections and infestations) | 3 | 1 | 1
COVID-19 pneumonia (Infections and infestations) | 1 | 0 | 0
Kidney Infection (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0
Carotid artery insufficiency (Nervous system disorders) | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0
Encephalopathy (Nervous system disorders) | 1 | 0 | 0
Hepatic encephalopathy (Nervous system disorders) | 0 | 0 | 1
Hypersensitive encephalopathy (Nervous system disorders) | 1 | 0 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0
Seizure (Nervous system disorders) | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0
Intra-abdominal hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Arrythmia (Cardiac disorders) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0
Cardiac tamponade (Cardiac disorders) | 0 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1 | 0
Anemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1 | 0
Liver function test increase (Investigations) | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=36) | Cohort 2 (N=11) | Cohort 3 (N=7)
Diarrhea (Gastrointestinal disorders) | 23 | 4 | 1
Nausea (Gastrointestinal disorders) | 17 | 1 | 2
Abdominal pain upper (Gastrointestinal disorders) | 7 | 2 | 1
Vomiting (Gastrointestinal disorders) | 6 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 6 | 1 | 0
Constipation (Gastrointestinal disorders) | 6 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 4 | 1 | 0
Fatigue (General disorders) | 20 | 4 | 3
Pyrexia (General disorders) | 2 | 3 | 2
Non-cardiac chest pain (General disorders) | 4 | 2 | 0
Peripheral edema (General disorders) | 4 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 6 | 3 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 | 2 | 3
Rash (Skin and subcutaneous tissue disorders) | 6 | 2 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 3 | 3 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 3 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 6 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 2 | 1
Hypokalemia (Metabolism and nutrition disorders) | 9 | 2 | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 8 | 4 | 1
Decreased appetite (Metabolism and nutrition disorders) | 10 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 2
Headache (Nervous system disorders) | 9 | 6 | 1
Dizziness (Nervous system disorders) | 7 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2022-09-21): https://cdn.clinicaltrials.gov/large-docs/10/NCT04383210/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-11): https://cdn.clinicaltrials.gov/large-docs/10/NCT04383210/SAP_001.pdf